CLINICAL TRIAL: NCT05092893
Title: Social Skills in Children With Developmental Coordination Disorder (DCD): a Cross-sectional Study
Brief Title: Social Skills in Children With Developmental Coordination Disorder (DCD)
Acronym: Social_DCD
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: b6702021000688
Record Dates: First submitted 2021-08-26; First posted 2021-10-26 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2021-08

CONDITIONS: Developmental Coordination Disorder
Keywords: Children; Social communication
MeSH Terms: conditions — Motor Skills Disorders; Communication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Developmental Coordination Disorder: INCLUSION:
  * Confirmed diagnosis of DCD
  * Comorbidities are allowed (f.e. ASD, ADHD, ADD,…)
  EXCLUSION:
  o Any other neurodevelopmental disorder which might affect motor development (f.e. CP).
  Interventions: Other: Online parental questionnaires

INTERVENTIONS:
Other: Online parental questionnaires — The SRS-2 is a parental 65-item questionnaire to detect difficulties in social responsiveness in children with autism spectrum disorder. Four different forms are available: preschoolers (2.5-4.5 years), school-aged children (4-18 years), adults (≥ 19 years) and adults self-report. In this study, only the form for school-aged children will be used.
  The DCDQ'07 is a parental 15-item questionnaire to detect the risk of DCD in children between 5 and 15 years of age. Parents are asked to compare their child's motor performance to his/her peers using a 5-point Likert scale. The total sum score is compared to age-specific cut-off scores to determine the risk of DCD. Belgian norms are available since 2007.

SUMMARY:
In this study we will examine the social-communicative skills of children with Developmental Coordination Disorder (DCD) by using online parental questionnaires in children aged 5 to 15y.

DETAILED DESCRIPTION:
Developmental Coordination Disorder (DCD) is a neurodevelopmental disorder described in the DSM-V characterized by motor coordination problems which significantly interfere with daily living activities and participation. The problems cannot be explained by another disorder and are already present in early life.

Although DCD is a 'motor' disorder, other domains may equally be affected. Children with DCD show lower health-related quality of life, more socio-emotional problems, and experience more academic difficulties. It has been proposed that social skills may mediate the emergence of socio-emotional problems at a later age. Previous research has suggested that socials skills of children with DCD may be altered. However, the process remains unclear. One possible hypothesis is that early motor coordination problems leads to avoiding or inhibits age-appropriate physical and social activities, which may reduce the opportunities to develop adequate socials skills and/or may impact negatively on a child's developing self-esteem and create a sense of isolation and exclusion.

Indeed, it has been reported that these children spend more time playing alone and are often onlookers instead of actively engaging in play. In general they exhibit a lower participation rate which may contribute to the reported poorer peer relations, less (deep) friendships, and a tendency for more bullying and loneliness. They also feel less competent in peer and social relations. Poorer social interaction skills and more social communication problems have been recognized in these children even interfering in non-verbal skills such as poorer recognizing of facial expressions and emotions and a reduced tendency to follow gaze which may be similar to children with ASD.

It can be debated if these social problems are comorbid or rather a secondary consequence.

With this study the investigators aim to map social responsiveness problems in children with Developmental Coordination Disorder and clarify if and which domains are most affected. The investigators defined the following research question: "Do children with Developmental Coordination Disorder experience social responsiveness problems compared to typically developing children? If so, which domains are most affected?".

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of DCD
* Comorbidities are allowed (f.e. ASD, ADHD, ADD,…)

Exclusion Criteria:

- Any other neurodevelopmental disorder which might affect motor development (f.e. CP).

Ages: 5 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: All children diagnosed with DCD in Belgium and The Netherlands between 5 and 15y.
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Social Responsiveness Questionnaire | through study completion, an average of 6 months
  Outcomes are reported in a total score and five subscales (social awareness, social cognition, social communication, social motivation and restricted interests and repetitive behavior).

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Van de Velde, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Roubaix A, Roeyers H, Van Waelvelde H, Bar-On L. Social responsiveness in children with developmental coordination disorder. Braz J Phys Ther. 2024 Jan-Feb;28(1):100591. doi: 10.1016/j.bjpt.2024.100591. Epub 2024 Feb 9. PMID 38394720